CLINICAL TRIAL: NCT07351630
Title: Feasibility, Acceptability, and Program Evaluation of A Parent Group to Support Child and Family Well-being
Brief Title: Building Blocks for Child and Family Well-being
Acronym: BBFW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Heather Prime, Associate Profesor, York University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4745
Record Dates: First submitted 2025-11-27; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Parenting Skills; Family Well-being; Family Cohesion
Keywords: Program Evaluation; Family Systems; Feasibility Study; Parenting Intervention; Caregivers; Parents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Parent Skills Group Program (Experimental): Caregivers who take part in a 6-week group program on parenting skills
  Interventions: Behavioral: Building Blocks for Family Well-being

INTERVENTIONS:
Behavioral: Building Blocks for Family Well-being — BBFW is a 6-week brief virtual program that promotes experiential learning, provides individually tailored strategies, and builds a community of support for caregivers. The program provides an integrated understanding of the family context, and equips caregivers with tools to help families connect, problem-solve, cope with stress, and thrive. The following topics are covered over 6 weeks: Introduction to the model; Getting to Know Your Family Members (e.g., temperament); Supporting Child Emotions; Promoting Positive Behaviours; Limit-Setting and Sibling Dynamics; Parenting Teams and Wrap-Up.

SUMMARY:
Background. Understanding emotions, stress, and conflicts within the family context is critical for promoting positive change. However, most support services for families often address child development, parenting, couple relationships separately without considering these as interacting systems that contributes to overall family well-being. This project is to evaluate an existing clinical service in York University Psychology Clinic (YUPC), "Building Blocks for Child and Family Well-being" (BBFW), which provides an integrated understanding of the family context, and equips caregivers with tools to help families connect, problem-solve, cope with stress, and thrive. BBFW is a brief virtual program that promotes experiential learning, provides individually tailored strategies, and builds a community of support for caregivers. The current study aims to examine the feasibility, acceptability, and effectiveness of the BBFW program within the York University Psychology Clinic (YUPC), with four objectives:

1. Evaluating the feasibility of implementing the BBWF program into YUPC clinical services, represented by enrolment rates, sample characteristics, retention (i.e., number of sessions attended, % dropout), adherence (i.e., completing in- and out-of-session activities), as well as the acceptability of the program among participants.
2. Examining sample and clinical characteristics of those attending the BBFW service
3. Exploring the effectiveness of the BBFW program through changes in family functioning and meta-emotion philosophy from pre- to post-intervention, as well as changes at 1- and 3-month follow-ups.
4. Evaluating and refining the program quality using participant quantitative and qualitative feedback.

The BBFW program is based on the best evidence from developmental, family, and relationship science. It aims to support family mental health and well-being through a holistic and sustainable approach, viewing the family as a set of multiple, interdependent systems. This program provides a brief, cost-effective, and accessible alternative with the potential to reduce the burden on traditional mental health and support services for Canadian families.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers aged 18 years or older participating in the BBFW program at York Univeristy's Psychology Clinic in Toronto, Ontario, Canada.
* Caregivers with children 18 years old or under are eligible to participate in the BBFW program.
* Caregivers must be residing in Ontario at the time of their service.
* Caregivers must also have access to a digital device with a screen (e.g., phone, tablet, computer) that can be used for virtual services.

Exclusion Criteria:

* Caregivers who do not consent to participate in research.
* Caregivers whose children are older than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Participants Enrolled Per month | Week 0
  Number of participants enrolled per month.
Geographic Reach | Week 0
  Cities/towns in Ontario families accessing the program reside. Data will be collected through the demographic questionnaire administered at baseline.
Retention | Week 0 to Week 18
  The percentage of participants who remain in study until the end of the follow up session.
Adherence | Week 1 to Week 6
  Number of sessions attended.
Adherence | Week 6
  Completion rate of in session activities.
Child Age Groups | Week 0
  Mean age of child of the parent who is seeking service. Data will be collected through the demographic questionnaire administered at baseline.
Primary Presenting Concern | Week 0
  Primary presenting concern of parent who is seeking service, collected at baseline using demographic questionnaire. Options include: child emotion regulation; child behavioural problems; challenging siblings dynamics; challenging co-parenting dynamics (working as a team with second parent); family stress, chaos, and/or conflict; other [please specify].
Family Clinical Characteristics | Week 2
  Family Clinical Characteristics include parent relationship dimension. The Relationship Dimension Scale (Lafrance, Henderson, & Mayman, 2020) is a 14-item tool for parents to reflect on different aspect of their relationships with their child/children. This is a qualitative measure that will be examined for themes arising in participating caregivers.
Family Clinical Characteristics | Week 1
  Family Clinical Characteristics include parent stress. The Family Stress Checklist includes 35 items which measures a parent's level of stress in 7 areas (i.e., financial, professional, physical, relational, environmental, child, parenting, discrimination). Each item is rated on a 5-item scale. Mean of items in each area will be calculated, with minimum score=1, maximum score=5. Higher scores correspond to higher level of stress in each area.
Client Satisfaction | Week 1, Week 2, Week 3, Week 4, Week 5, Week 6
  Client Satisfaction will be measured using surveys and participant qualitative feedback. A brief satisfaction survey will be administered weekly at the end of each group session. This survey consists of 4 questions about the content, facilitation, group activities/discussion, as well as an open-ended question for general feedback about the session. In the end, participant will be asked to complete another satisfaction survey about the program overall. Means of the survey items will be calculated. Minimum score=1, maximum score=4. Higher scores correspond to higher satisfaction.
Client Acceptability | Week 6
  Percentage of participants reporting at least 'good' on 80 % or more indicators on an Implementation Acceptability Scale that will assess attitude, burden, perceived effectiveness, and ethicality. Minimum score=7, maximum score=35. Higher scores correspond to better outcomes.

SECONDARY OUTCOMES:
Pre-Post Change in Parent Reported Family Functioning | Changes from Week 0 to Week 6; from Week 0 to Week 10; from Week 0 to Week 18
  Changes in Family Functioning will be assessed using the McMaster Family Assessment Device (FAD; Epstein et al., 1983). The scale has 60 items representing 7 subscales: Problem Solving, Communication, Roles, Affective Responsiveness, Affective Involvement, Behavior Control, General Functioning. Each item is rated on 4 point scale. Mean of each subscale will be calculated. For each subscale, minimum score=1, maximum score=4. Higher scores correspond to worse outcomes (i.e., less healthy family functioning).
Pre-Post Change in Parent Meta-Emotion Philosophy | Changes from Week 0 to Week 6; from Week 0 to Week 10; from Week 0 to Week 18
  Changes in Parent Meta-Emotion Philosophy will be assessed using the Emotion-Related Parenting Styles Scale-Short Form (ERPS-SF; Paterson et al., 2012).
  The scale has 20 items, each rated on a 5-point Likert Scale. Mean of items representing 4 parenting styles will be calculated. For each parenting style, minimum score=1, maximum score=5. The style with highest average score indicates the participant's emotion-related parenting style.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Prime, PhD, Principal Investigator — York University
Locations (2):
- Canada (2):
  - York University,, Toronto, Ontario
  - York University Psychology Clinic, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Philipp DA, Prime H, Darwiche J. An ultra-brief systemic intervention to address child mental health symptomatology. Fam Process. 2023 Jun;62(2):469-482. doi: 10.1111/famp.12875. Epub 2023 Mar 23. PMID 36959726
- [Background] Lafrance, A., Henderson, K. A., & Mayman, S. (2020). Emotion-focused family therapy: A transdiagnostic model for caregiver-focused interventions. American Psychological Association
- [Background] Dishion TJ, Shaw D, Connell A, Gardner F, Weaver C, Wilson M. The family check-up with high-risk indigent families: preventing problem behavior by increasing parents' positive behavior support in early childhood. Child Dev. 2008 Sep-Oct;79(5):1395-414. doi: 10.1111/j.1467-8624.2008.01195.x. PMID 18826532
- [Background] Bennett T, Georgiades K, Gonzalez A, Janus M, Lipman E, Pires P, Prime H, Duku E, Jambon M, McLennan JD, Gross J; Making the Race Fair Study Team. Targeted Child Mental Health Prevention and Parenting Support Within a Canadian Context: A Randomized Controlled Trial Evaluating the U.S.-Developed Family Check-Up(R). Prev Sci. 2025 May;26(4):555-567. doi: 10.1007/s11121-024-01741-3. Epub 2024 Nov 22. PMID 39572487